CLINICAL TRIAL: NCT01578200
Title: Outcome Study of Lanthanum Carbonate Compared With Calcium Carbonate on Cardiovascular Mortality and Morbidity in Patients With Chronic Kidney Disease on Hemodialysis (CKD5D)
Brief Title: Outcome Study of Lanthanum Carbonate Compared With Calcium Carbonate in Hemodialysis Patients : Landmark Study
Acronym: LANDMARK
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Collaborators: Showa University School of Medicine (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRIGU1111; UMIN000006815 (Registry Identifier: UMIN Clinical Trials Registry)
Record Dates: First submitted 2012-04-13; First posted 2012-04-16 (Estimated); Last update posted 2020-11-30 (Actual); Status verified 2019-03

CONDITIONS: Hemodialysis; Hyperphosphatemia
Keywords: CKD-MBD; phosphate-binder; vascular calcification; mortality; dialysis; Hemodialysis patients with hyperphosphatemia
MeSH Terms: conditions — Hyperphosphatemia; Chronic Kidney Disease-Mineral and Bone Disorder; Vascular Calcification | interventions — lanthanum carbonate; Calcium Carbonate

ARMS (2):
- Lanthanum carbonate (Experimental): Patients are given Lanthanum Carbonate oral administration after meals three times per day in total daily dose of 750-2250mg.
  Interventions: Drug: Lanthanum Carbonate
- Calcium Carbonate (Active Comparator): Patients are given Calcium carbonate oral administration after meals three times per day in total daily dose of 3.0g.
  Interventions: Drug: Calcium Carbonate

INTERVENTIONS:
Drug: Lanthanum Carbonate
  Arms: Lanthanum carbonate
Drug: Calcium Carbonate
  Arms: Calcium Carbonate

SUMMARY:
The purpose of this study is to demonstrate decrease in cardiovascular mortality and morbidity in Japanese hemodialysis patients treated with Lanthanum carbonate compared with those with Calcium carbonate.

DETAILED DESCRIPTION:
Elevated serum phosphate and calcium in dialysis patients are independently associated with increased risk of arterial calcification and mortality. Calcium-based phosphate binders can induce hypercalcaemia and are associated with progression of vascular calcification. A recent randomized study demonstrated that sevelamer, a non-calcium-based phosphate binders, reduced mortality in elderly hemodialysis patients compared with calcium-based phosphate binders. Lanthanum carbonate is another efficacious and well-tolerated non-calcium phosphate binder. A post-hoc survival analysis of lanthanum carbonate versus standard therapy suggested a survival benefit of lanthanum carbonate treatment for elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* hemodialysis patients with hyperphosphatemia who require phosphate binders
* hemodialysis for more than 3 months
* patients who have at least one calcification risk factor (elderly > 65 years, postmenopausal woman, type 2 diabetes mellitus)
* intact-PTH < or = 240pg/mL
* life expectancy > 1 year
* with written informed consent

Exclusion Criteria:

* contraindications to lanthanum carbonate and calcium carbonate
* swallowing disorders
* severe GI disorders
* history of obstructed bowels
* history of IHD/stroke within 6 months before randomization
* NYHA classification Ⅲ-Ⅳ
* severe liver dysfunction (AST or ALT greater than 3 times the upper limit of institution
* require treatment of arrhythmia
* severe malnutrition
* malignancy of any type within the last five years
* peritoneal dialysis patients
* pregnant or possibly pregnant women or women on lactation and planned to get pregnant within study term
* ineligible patients according to the investigator's judgment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2309 (Actual)
Dates: Start 2011-12-24; Primary Completion 2019-03-25 (Actual); Study Completion 2019-03-25 (Actual)

PRIMARY OUTCOMES:
Cardiovascular event free survival time. | 3 years
  Cardiovascular event consisting of
  1. death due to cardiovascular diseases including sudden cardiac death (ICD-10 codes R96.0/96.1),
  2. nonfatal myocardial infarction,
  3. nonfatal cerebral stroke including transient ischemic attack, TIA,
  4. unstable angina,
  5. hospitalization for heart failure,
  6. hospitalization for ventricular arrhythmia

SECONDARY OUTCOMES:
Overall survival | 3 years
Secondary hyperparathyroidism free survival | 3 years
Hip fracture free survival | 3 years
Quality of life questionnaire (KDQOL-SF, v1.3) | 3 years
Bone mineral density (DEXA) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Tadao Akizawa, MD, PhD, Principal Investigator — Showa University
Locations (1):
- Showa University, Shinagawa, Tokyo, Japan

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086
- [Derived] Ogata H, Fukagawa M, Hirakata H, Kagimura T, Fukushima M, Akizawa T; LANDMARK Investigators and Committees. Effect of Treating Hyperphosphatemia With Lanthanum Carbonate vs Calcium Carbonate on Cardiovascular Events in Patients With Chronic Kidney Disease Undergoing Hemodialysis: The LANDMARK Randomized Clinical Trial. JAMA. 2021 May 18;325(19):1946-1954. doi: 10.1001/jama.2021.4807. PMID 34003226